CLINICAL TRIAL: NCT05310591
Title: Combination of an Anti-PD1 Antibody With Tisagenlecleucel Reinfusion in Children, Adolescents and Young Adults With Acute Lymphoblastic Leukemia After Loss of Persistence
Acronym: CAPTiRALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP200132
Record Dates: First submitted 2022-03-09; First posted 2022-04-05 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-02

CONDITIONS: B Acute Lymphoblastic Leukemia; Acute Lymphoblastic Leukemia, in Relapse
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with MRD negative disease status: Time to Event Continual Reassessment Method (TITE-CRM) (Experimental)
  Interventions: Drug: Decreasing starting times for beginning nivolumab (Time to Event Continual Reassessment Method (TITE-CRM) )
- For relapsed patients (Experimental)
  Interventions: Drug: Nivolumab starting at day -1

INTERVENTIONS:
Drug: Decreasing starting times for beginning nivolumab (Time to Event Continual Reassessment Method (TITE-CRM) ) — Patients included first receive a lympho-depleting chemotherapy by Fludarabine / Cyclophosphamide. tisagenlecleucel infusion should then be administered 2 to 14 days after completion of chemotherapy.
  Nivolumab (Opdivo®) will be given intravenously at 3mg/kg every 2 weeks. It will include patients with MRD negative disease status.
  1. Four decreasing starting times for beginning nivolumab (day 14, day 11, day 5 and day -1) will be available for testing
  2. Patients will be enrolled sequentially by cohorts of 3 with escalation between cohorts based only on the limiting toxicities between infusion and D28
  Nivolumab will be given until 12 months after tisagenlecleucel infusion in case of response.
  Arms: Patients with MRD negative disease status: Time to Event Continual Reassessment Method (TITE-CRM)
Drug: Nivolumab starting at day -1 — It will include relapsed patients. Patients included first receive a lympho-depleting chemotherapy by Fludarabine / Cyclophosphamide. tisagenlecleucel infusion should then be administered 2 to 14 days after completion of chemotherapy.
  Nivolumab (Opdivo®) will be given intravenously at 3mg/kg every 2 weeks.
  -nivolumab starting at day -1.
  Nivolumab will be given until 12 months after tisagenlecleucel infusion in case of response.
  Arms: For relapsed patients

SUMMARY:
Tisagenlecleucel (CTL019) is an anti-CD19 autologous Chimeric Antigen Receptor (CAR) T-cell therapy, which has shown dramatic early results in advanced ALLs. Early loss of B-cell aplasia (recovery of B-cells in marrow/ peripheral blood within 6 months after infusion), a marker of the loss or non-functionality of the CAR T-cells, is associated to a very high risk of relapse. A reinfusion of CTL019, even after Fludarabine-Cyclophosphamide reconditioning, frequently fails to induce further expansion as observed in UPENN studies and in the Robert Debré Hospital experience.

Non-persistence of CAR T-cells may be due to immune- mediated rejection or environment-mediated suppression of their growth. Evidence for increased PD-1 expression in CAR T-cells between infusion and peak expansion has been demonstrated in clinical samples.

Preclinical data and few clinical data support a role of PD- 1-PD-L1 blockade in improving the effectiveness of CAR T-cell therapy.

The objectives of this phase I/II study is to determine the safety, efficacy and feasibility of Nivolumab (Opdivo®)- an anti-PD1 treatment- combined to tisagenlecleucel in a cohort of relapsed or refractory B-ALL patients, aged 1-25 years old, previously treated by tisagenlecleucel (Kymriah®), with a demonstrated early loss of B-cell aplasia (within 6 months), a surrogate marker of the loss of CAR T-cells or their non- functionality.

More specifically, the main objectives are:

• In cohort 1 that includes patients with a MRD negative disease status combined to an early loss (within 6 months) of B-cell aplasia :

To determine the optimal starting time of Nivolumab (Opdivo®) in terms of safety and efficacy among 4 candidate time points (day 14, day 11, day 5, and day - 1).

• In cohort 2 that includes relapsed patients with an early loss (within 6 months) of B-cell aplasia :

To estimate the feasibility in terms of safety and efficacy of a very early start of nivolumab (day-1), prior to the reinfusion of tisagenlecleucel

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 1 to 25 years (pediatric and young adults) with a history of CD19+ relapsed or refractory B-ALL (any relapse after HSCT, 2nd relapse or later, refractory ALL).
* Patient must have a second tisagenlecleucel (Kymriah ®) product available
* Cohort 1: previously treated by tisagenlecleucel (Kymriah ®), and who present an early loss of B-cell aplasia defined by blood B lymphocytes < 10 /mm3 and/ or < 3% of total lymphocytes (< 6 months after infusion) while still being in CR with undetectable MRD
* Cohort 2: previously treated by tisagenlecleucel (Kymriah ®), who present a loss of B-cell aplasia defined by blood B lymphocytes < 10 /mm3 and/ or < 3% of total lymphocytes and a CD19+ ALL detectable disease in the marrow and/or Blood
* Life expectancy > 12 weeks.
* Karnofsky (age > 16) Lansky (age < 16) > 70 at screening.
* No organ dysfunction
* Who have signed an informed consent
* Affiliation to social security or any health insurance (as a beneficiary or assignee)

Exclusion Criteria:

* Patient has received intervening therapy for leukemia after first tisagenlecleucel infusion (chemotherapy, anti leukemic immunotherapy, ITK, allogeneic HSCT).
* Patient has an active autoimmune disease requiring systemic treatment within the past 2 years.
* Patient has known history of, or any evidence of active, non-infectious pneumonitis.
* Patient has a history of non-infectious pneumonitis that required steroid or has current pneumonitis.
* Had receive prior therapy with an anti-PD1, Anti- PDL1 or anti-PDL2 agent.
* Patient has hypersensivity to pembrolizumab/ nivolumab or one of its excipients
* Patient has received a live vaccine injection within 45 days of planned start of study therapy.
* Patients with concomitant genetic syndromes associated with bone marrow failure states: such as patients with Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome. Patients with Down syndrome will not be excluded.
* Patients with Burkitt's lymphoma/leukemia
* Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease.
* Prior treatment with any gene therapy product except first tisagenlecleucel (Kymriah ®) injection.
* Prior treatment with any anti-CD19/anti-CD3 therapy, or any other anti-CD19 therapy, except for patients pre-treated with blinatumomab and/or tisagenlecleucel (Kymriah®)
* Prior anti-cancer monoclonal antibody within 4 weeks before starting the study.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade1 or at baseline) from adverse events due to a previously administered agent.
* Active or latent hepatitis B or active hepatitis C (test within 8 weeks of Screening), or any uncontrolled infection at Screening.
* Human immunodeficiency virus (HIV) positive test within 8 weeks of Screening.
* Presence of grade 2 to 4 acute or extensive chronic GVHD.
* Active CNS involvement by malignancy, defined as CNS-3 per NCCN guidelines. Note: Patients with history of CNS disease that has been effectively treated will be eligible.
* Uncontrolled acute life threatening bacterial, viral or fungal infection at Screening.
* Previous or concurrent malignancy with the following exceptions:

  * Adequately treated basal cell or squamous cell carcinoma
  * in situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to the study.
  * A primary malignancy completely resected and in CR for ≥ 5 years
* Pregnant or lactating women (female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion)
* Patient with hypersensivity to Fludarabine and/or cyclophosphamide and/or tisagenlecleucel and/or nivolumab or one of their excipients.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with limiting-toxicities | at day 28
  Limiting toxicities are defined by the occurrence of either
  - Related to CAR-T cells infusion: CRS or aGVH: limiting toxicity will be defined as toxicity ≥ 4 ICANs: limiting toxicity will be defined as toxicity ≥ 3 (excepted grade 3 seizure, ie focal, generalized seizure that resolves rapidly)
  - Related to nivolumab: immune related myocarditis, pneumonitis, encephalitis: limiting toxicity will be defined as toxicity ≥ 4
Efficacy assessed by Minimal residual disease (MRD) negative Complete remission (CR) and B cell aplasia. | at 3 months
  MRD negative CR is defined by undetectable disease at a 10-4 sensitivity threshold B cell aplasia is defined by blood B lymphocytes < 10 /mm3 and/or < 3% of total lymphocytes

SECONDARY OUTCOMES:
Incidence of B cell aplasia | at 6 months
Increase of B cell aplasia duration compared to the previous one observed | up to 24 months
Proportion of patients with Disease best response | up to three months
Proportion of patients with Complete remission | at 1 month
Proportion of patients with Complete remission | at 3 months
Proportion of patients with Complete remission | at 6 months
Proportion of patients with Complete remission | at 12 months
Proportion of patients with Minimal residual disease | at 1 month
Proportion of patients with Minimal residual disease | at 3 months
Proportion of patients with Minimal residual disease | at 6 months
Proportion of patients with Minimal residual disease | at 12 months
Overall survival | at one year
Overall survival | at 2 years
Event Free Survival (EFS) | at 1 year
Event Free Survival (EFS) | at 2 years
Incidence of Grade 3 adverse events | up to 2 years
Incidence of Grade 3, 4 or 5 nivolumab-related adverse events | up to 2 years
Incidence of GVHD | up to one year

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHRU Bordeaux, Bordeaux
  - CHRU Lille, Lille
  - HCL - Lyon Sud, Lyon
  - HCL, Lyon
  - Hôpital pour enfants - La Timone, Marseille
  - CHU Montpellier - Hopital Arnaud de Villeneuve, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes - Hopital Mère-enfants, Nantes
  - Robert Debre hospital, Paris
  - Saint Louis hospital, Paris
  - CHU Rouen, Rouen
  - CHRU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided